CLINICAL TRIAL: NCT00368524
Title: Cost Effective Treatment for Dually Diagnosed Homeless
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Penelope Baker Jester, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F920822004; 1R01DA011789 (NIH)
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2006-08

CONDITIONS: Cocaine Dependence; Mental Disorder; Homelessness; Unemployment
Keywords: cocaine dependence; mental disorder; dual diagnoses; homelessness
MeSH Terms: conditions — Cocaine-Related Disorders; Mental Disorders

INTERVENTIONS:
Behavioral: contingency management and behavioral day treatment

SUMMARY:
This randomized controlled trial examined whether an abbreviated treatment using abstinence contingency management for housing and work/training (CM, n=103) with cocaine dependent, non-psychotic, dually diagnosed homeless persons, would show non-inferior outcomes compared to the full treatment (CM+, n=103). It was hypothesized that CM+ would show superior abstinence and retention outcomes, but that CM, with components derived from previously effective behavioral day treatment, would obtain non-inferior outcomes, defined as 75% or more of those observed for the full treatment (CM+) during active treatment months 1-6. The CM+ included all CM components but added behavioral day treatment that included voucher reinforcement of $7.50-15.00, for objective weekly therapeutic goal attainment in five domains of functioning: drug dependence, homelessness, unemployment, non-drug related recreational activities, and behavioral, health, or mental health problems. Abstinence was assessed by observed urine specimen collection and weekly testing weeks 1-52, and randomly, bi-monthly for months 13-18. Abstinence, homelessness, employment and other outcomes were also assessed at baseline, 2, 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria: McKinney Act criteria for homelessness; DSM IV diagnosis for Cocaine Dependence; self-reported use within the last 2 weeks; psychological distress indicated by score of 70 on 1 or more Brief Symptom Inventory scales; willingness to participate; no plans to move from Birmingham area for 18 months;

-

Exclusion Criteria: cognitive impariment precluding informed consent; requiring immediate inpatient medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-11; Study Completion 2005-11

PRIMARY OUTCOMES:
abused drug abstinence measured by observed urine specimen testing weeks 1-52, and bimonthly months 13-18

SECONDARY OUTCOMES:
abstinence, housing, employment and other outcomes at 0, 2, 6, 12 and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse B. Milby, Ph.D. ABPP, Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Background] Milby JB, Schumacher JE, Wallace D, Freedman MJ, Vuchinich RE. To house or not to house: the effects of providing housing to homeless substance abusers in treatment. Am J Public Health. 2005 Jul;95(7):1259-65. doi: 10.2105/AJPH.2004.039743. PMID 15983278
- [Derived] Milby JB, Schumacher JE, Vuchinich RE, Freedman MJ, Kertesz S, Wallace D. Toward cost-effective initial care for substance-abusing homeless. J Subst Abuse Treat. 2008 Mar;34(2):180-91. doi: 10.1016/j.jsat.2007.03.003. Epub 2007 May 23. PMID 17512156